CLINICAL TRIAL: NCT06794190
Title: Characterization of Hepatopathy in Turner Syndrome: Analysis of Determinants in an Observational Study
Brief Title: Characterization of Hepatopathy in Turner Syndrome: Analysis of Determinants
Status: Recruiting | Type: Observational
Sponsor: IRCCS Azienda Ospedaliero-Universitaria di Bologna (Other)
Responsible Party: Sponsor
Other Study IDs: LIVER_TS-2023
Record Dates: First submitted 2024-12-30; First posted 2025-01-27 (Actual); Last update posted 2025-01-27 (Actual); Status verified 2024-12

CONDITIONS: Turner Syndrome
MeSH Terms: conditions — Turner Syndrome

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
The present study is therefore aimed at investigating the prevalence of hepatic alterations (laboratory and imaging) in adult patients with TS and generating hypothesissto the possible etiopathogenetic factors most involved, as well as evaluating the correlation between biochemical and structural abnormalities.

Thus, the study could provide relevant etiopathogenetic and prognostic results on the development of hepatopathy in TS patients.

DETAILED DESCRIPTION:
The study is an observational retrospective cohort type; patients with TS in longitudinal monitoring at the U.O.C. of Endocrinology and Diabetes Prevention and Care, DIMEC, of IRCCS Policlinico S. Orsola of Bologna will be enrolled. The diagnosis of TS was made for most patients by the Pediatrics unit of Policlinico S. Orsola; in rare cases it was performed in adulthood by our operating unit or at another center; in all cases, the diagnosis was made by karyotype analysis on peripheral blood.

The patients, as per clinical practice, underwent clinical evaluation with measurement of anthropometric parameters; an evaluation of the patients' medical history will be performed, paying attention to possible diagnosis of metabolic comorbidities and autoimmune diseases. Complete information regarding the history of menstrual cycles and replacement therapies used will also be collected. Finally, laboratory investigations are planned.

ELIGIBILITY:
Inclusion Criteria:

* Diagnosis of Turner syndrome made by karyotype analysis on peripheral blood.
* Age 18 years or older
* Written informed consent obtained

Exclusion Criteria:

* TS patients on therapy with drugs responsible for significant liver enzyme alterations (liver function alteration, LFA).

Min Age: 18 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Gender Based: Yes — * Diagnosis of Turner syndrome made by karyotype analysis on peripheral blood.
  * Age 18 years or older
  * Written informed consent obtained
Study Population: The study population will be enrolled from the cohort of adult TS patients under longitudinal monitoring at the U.O.C. of Endocrinology and Diabetes Prevention and Care IRCCS Policlinico S. Orsola.
Sampling Method: Non-Probability Sample
Enrollment: 120 (Estimated)
Dates: Start 2025-01-07 (Actual); Primary Completion 2026-01-06 (Estimated); Study Completion 2026-01-07 (Estimated)

PRIMARY OUTCOMES:
Factors associated with hepatopathy | Baseline
  Hepatopathy, defined as the presence of at least one of the following conditions:
  * AST ≥ 35 UI/L
  * ALT ≥ 35 UI/L
  * GGT ≥ 38 UI/L
  * ALP ≥ 116 UI/L
  * Presence of hepatic steatosis

SECONDARY OUTCOMES:
Comparison of liver morpho-functional parameters with results obtained by fibroscan. | Baseline
  Liver stiffness measurement (kPa)
Comparison of liver morpho-functional parameters with results obtained by fibroscan. | Baseline
  Spleen stiffnes measurement (kPa)

CONTACTS AND LOCATIONS:
Overall Officials: Alessandra Gambineri, MD, Principal Investigator — IRCCS Azienda Ospedaliero-Universitaria di Bologna
Locations (1):
- IRCCS Azienda Ospedaliero-Universitaria di Bologna, Bologna, Italy

IPD SHARING:
Plan to Share IPD: No